CLINICAL TRIAL: NCT01020981
Title: National Guard Outreach and Linkage to Treatment
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: RRP 09-420
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: PTSD; Depression; Reintegration; Veterans Health
Keywords: OEF/OIF; Peer Group; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Michigan State Army National Guard soldiers who have returned from OEF/OIF deployments starting December 2008
- Group 2: Indiana State Army National Guard soldiers who have returned from OEF/OIF deployments starting December 2008

SUMMARY:
This project will add an evaluation/research component to an existing peer outreach program, now implemented for over 1100 soldiers in the Michigan Army National Guard. Preliminary work will be completed in three areas. We will conduct semi-structured interviews with soldiers, Buddies, and National Guard leadership and develop and pilot test survey items relevant to implementation. Further, we will develop and pretest survey items relevant to determining soldier symptomatic and functional status. We will also conduct a small feasibility study, fielding the newly developed survey to a representative sample of recently returned National Guard members from Michigan and Indiana, to determine response rates and veteran willingness to allow access to linkable PDHA/PDHRA data and health services data. Finally, we will construct a merged, de-identified longitudinal dataset comprised of Post-Deployment Health Assessment and Reassessment data, Military Health System/TRICARE, and VA services data from National Guard soldiers in Michigan and comparison states of Indiana and Ohio. This will allow a longitudinal assessment of services initiation and retention for the entire Guard populations in these states.

DETAILED DESCRIPTION:
Background:

Soldiers returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) commonly experience symptoms of PTSD, depressive disorders, and interpersonal difficulties. Forty-two percent of National Guard (NG) soldiers report symptoms suggesting a need for evaluation. Unfortunately, only half with mental health needs initiate treatment in the VA or elsewhere. Stigma remains an important barrier. Proactive peer outreach may successfully address stigma and facilitate appropriate treatment use. In the recently implemented Michigan Guard Buddy*to*Buddy (B2B) program, all returning MIARNG soldiers are assigned a first-tier "Buddy" from their unit who systematically telephones them to "check in" regarding key areas of functioning and symptoms. Soldiers may also be referred to second-tier Buddies, veterans outside the Guard trained in motivational interviewing and supervised by professional staff. The goal of the program is to identify soldiers in need of evaluation and connect them to care in a timely fashion.

We will conduct preliminary work that will allow us to assess the need for and the feasibility of adding a rigorous evaluation/research component to the B2B program.

Objectives:

The goal of this RRP is to assess the need for AND the feasibility of a larger VA study that would use a strong quasi-experimental design (time series analysis with comparison groups) to examine the impact of the B2B program on returning NG veteran mental health treatment initiation, retention, symptoms, and functional outcomes.

Specific RRP aims are to:

1. Prepare for and initiate a formative evaluation of the Buddy*to*Buddy program in the Michigan Army National Guard (MI ARNG).
2. Develop and determine the feasibility of a confidential surveys for National Guard veterans in Michigan and Indiana that elicit information regarding B2B processes (in MI ARNG), VA outreach processes, mental health symptoms, substance use, and treatment initiation and retention.
3. Construct a de-identified linked dataset consisting of PDHA/PDHRA data, Military Treatment Facility/TRICARE service provider use, and VA service use for MI ARNG and NG soldiers in contiguous states of Indiana and Ohio. Conduct preliminary analyses of these data.

Methods:

Preliminary work will be completed in two areas. We will begin a formative evaluation of the implementation of the B2B program, using an augmented qualitative RE-AIM Plus framework, multiple data sources and data collection techniques, and conducting field observations and interviews with program stakeholders. Personnel at all levels, including NG leadership, Buddies, and soldiers, will be part of this process.

We will also develop and refine survey items relevant to understanding B2B implementation and soldier symptom and functional status. We will test procedures for fielding this survey in Michigan and a comparison state, assessing response rates, and using data to inform the design of a larger study of soldier outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Returning MI ARNG member participating in the Buddy-to-Buddy program

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MI, IN, and OH ARNG
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia T. Valenstein, MD AB, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Valenstein M, Gorman L, Blow AJ, Ganoczy D, Walters H, Kees M, Pfeiffer PN, Kim HM, Lagrou R, Wadsworth SM, Rauch SA, Dalack GW. Reported barriers to mental health care in three samples of U.S. Army National Guard soldiers at three time points. J Trauma Stress. 2014 Aug;27(4):406-14. doi: 10.1002/jts.21942. PMID 25158634
- [Result] Burnett-Zeigler I, Valenstein M, Ilgen M, Blow AJ, Gorman LA, Zivin K. Civilian employment among recently returning Afghanistan and Iraq National Guard veterans. Mil Med. 2011 Jun;176(6):639-46. doi: 10.7205/milmed-d-10-00450. PMID 21702380
- [Result] Burnett-Zeigler I, Ilgen M, Valenstein M, Zivin K, Gorman L, Blow A, Duffy S, Chermack S. Prevalence and correlates of alcohol misuse among returning Afghanistan and Iraq veterans. Addict Behav. 2011 Aug;36(8):801-6. doi: 10.1016/j.addbeh.2010.12.032. Epub 2011 Jan 13. PMID 21482030
- [Result] Dalack GW, Blow AJ, Valenstein M, Gorman L, Spinner J, Marcus S, Kees M, McDonough S, Greden JF, Ames B, Francisco B, Anderson JR, Bartolacci J, Lagrou R. Public-academic partnerships: working together to meet the needs of Army National Guard soldiers: an academic-military partnership. Psychiatr Serv. 2010 Nov;61(11):1069-71. doi: 10.1176/ps.2010.61.11.1069. PMID 21041342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interview and focus group participants and survey pre-testers participated during drill weekends in November and December 2010. Surveys were mailed to MI NG members in March 2011 with 2nd mailing in April 2011, and 3rd mailing in May 2011 and to Indiana NG members with first mailing in Sept 2011 , 2nd in Oct 2011, and 3rd mailing in Nov 2011.
Pre-assignment Details: Fifteen soldiers in Michigan participated in interviews or focus groups during survey development. The survey was fielded to 300 Soldiers, 150 in Michigan and 150 in Indiana. A total of 141 Soldiers either returned a survey and/or completed an interview and were considered enrolled in the study. This is detailed in Participant Flow.
Groups:
- Michigan Army National Guard: Michigan Army National Guard soldiers who have returned from OEF/OIF deployments starting December 2008
- Indiana Army National Guard: Indiana State Army National Guard soldiers who have returned from OEF/OIF deployments starting December 2008
Period: Overall Study
Arm/Group | Michigan Army National Guard | Indiana Army National Guard
Started | 150 | 150
Completed | 66 | 60
Not Completed | 84 | 90
Not completed — Did not return mailed survey | 74 | 58
Not completed — Survey returned undeliverable | 8 | 32
Not completed — Participant declined to complete survey | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Michigan Army National Guard: Michigan State Army National Guard soldiers who have returned from OEF/OIF deployments starting December 2008
- Total: Total of all reporting groups
Arm/Group | Michigan Army National Guard | Indiana Army National Guard | Total
Number analyzed (Participants) | 81 | 60 | 141
Age, Customized [Number; unit: participants]
  18-21 yrs | 5 | 0 | 5
  22-30 yrs | 23 | 9 | 32
  31-40 yrs | 15 | 8 | 23
  41-50 yrs | 18 | 28 | 46
  >50 yrs | 3 | 15 | 18
  Unknown | 17 | 0 | 17
Sex/Gender, Customized [Number; unit: participants]
  Male | 60 | 46 | 106
  Female | 3 | 10 | 13
  Unknown | 18 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Feasibility-response Rate
Description: Response rate of Soldiers to a mailed survey.
Time Frame: Survey was fielded to Michigan National Guard Service Members on three occasions, March 2011, April 2011, and May 2011. The survey was also fielded to Indiana National Guard Service Members on September 2011, October 2011, and November 2011.
Population: 8 or 5% of surveys to Michigan NG Soldiers were not deliverable. 32 (21%) of Indiana NG soldier surveys were not deliverable.
  66 of 142 delivered surveys to MI soldiers were returned for a response rate of 46%. 60 of 118 deliverable surveys to Indiana NG Soldiers were returned for a response rate of 51%.
Measure: Number; unit: % of Soldiers returning mailed survey
Groups:
- Indiana Army National Guard: Indiana Army National Guard soldiers who have returned from OEF/OIF deployments starting December 2008
Arm/Group | Michigan Army National Guard | Indiana Army National Guard
Number analyzed (Participants) | 142 | 118
% of Soldiers returning mailed survey | 46 | 51

2. Secondary Outcome: Depressive Symptoms
Description: The 21-item Beck Depression Inventory-2nd Edition (BDI-II) was used to assess depressive symptoms. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Survey was fielded to MIARNG in March 2011 (INARNG in September 2011). Soldiers who did not respond were sent two additional mailings with surveys in April 2011(INANG-October 2011) and May 2011 (INANG-November 2011).
Population: Data were analyzed for those with complete outcome data. Thus, 1 participant in Michigan Army National Guard and 1 participant in Indiana Army National Guard are not included in these results.
Measure: Mean (Standard Deviation); unit: units on a BDI-II scale
Groups:
- Michigan Army National Guard: Michigan State Army National Guard soldiers who have returned from OEF/OIF deployments after December 2008
- Indiana Army National Guard: Indiana State Army National Guard soldiers who have returned from OEF/OIF deployments after December 2008
Arm/Group | Michigan Army National Guard | Indiana Army National Guard
Number analyzed (Participants) | 65 | 59
units on a BDI-II scale | 5.01 (6.02) | 4.81 (5.81)

3. Secondary Outcome: PTSD Symptoms
Description: The PCL is a 17-item self-report checklist of PTSD symptoms based closely on the DSM-IV criteria. The PCL-M is a military version and questions refer to "a stressful military experience". Total possible scores range from 17 to 85. Higher scores indicate more symptoms of PTSD and a cut-off score of 50 is used for indicating a probable diagnosis of combat-related PTSD.
Time Frame: as for outcome 2
Population: 86% of MI NG soldiers who completed surveys returned a complete PCL scale and 87% of IN NG soldiers who completed surveys returned a complete PCL scale.
Measure: Mean (Standard Deviation); unit: units on PCL scale
Arm/Group | Michigan Army National Guard | Indiana Army National Guard
Number analyzed (Participants) | 57 | 52
units on PCL scale | 31.61 (15.88) | 29.56 (15.80)

ADVERSE EVENTS:
Time Frame: Two months, November and December 2010
Arm/Group | Michigan Army National Guard | Indiana Army National Guard
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/60
Other Adverse Events (participants affected / at risk) | 0/81 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes